CLINICAL TRIAL: NCT06404632
Title: A Group Intervention for Promoting Health-related Habits in Individuals With Disabilities (LEV-G)
Brief Title: A Group Intervention for Promoting Health-related Habits (LEV-G)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other); Promobilia Foundation (Other)
Responsible Party: Principal Investigator, Douglas Sjowall, PhD, Associate professor, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: The LEV Project (group)
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Life Style; Health-Related Behavior; Disabilities Mental; Disability Physical; Acceptability of Health Care
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Feasibility trial with pre, peri, post and follow-up measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lev-g (group intervention) (Experimental): Lev-g includes three sessions + a booster session using psychoeducation, motivational interviewing, and applied behavioral analyses. Lev-g is done in groups to enable support and tips from others. There is no control condition. Only one arm to test feasibility.
  Interventions: Behavioral: Lev-g

INTERVENTIONS:
Behavioral: Lev-g — Lev-g includes three sessions + a booster session using psychoeducation, motivational interviewing, and applied behavioral analyses. Lev-g is done in groups to enable support and tips from others.

SUMMARY:
Health-related habits influences mental and physical health. Still, treatment of health-related habits, which can help to remedy health problems, is often not done at all or very superficially. Multiple guidelines emphasize the importance of prioritizing health-related habits, but there is a lack of implemented models. To solve this, the investigators have developed a transdiagnostic, interprofessional material intended for several care settings. The Lev-g intervention is intended for groups. There is also an individual version of Lev that has its on registration in Clinical Trails.

DETAILED DESCRIPTION:
Lev is a brief, transdiagnostic, interprofessional intervention targeting health-related habits that is intended for several care settings. The main population intended is individuals with neurodevelopmental disorders or parents or close relations to children with disabilities. This study will therefore be open for participants recruited from several types of healthcare services in Sweden.

Study 1: The feasibility trial investigates the following questions:

Completion: How many participants that started Lev completed the intervention? What were the reasons for not not completing Lev? How many sessions did the participants complete? Lev includes screening (Lev-s), three sessions + one booster session.

Level of acceptability: Was Lev perceived as creditable and satisfactory by healthcare workers and participants? Treatment credibility will be measured before Lev and after the last session for both participants and healthcare workers. Treatment satisfaction will be evaluated after each session and after the intervention is completed. Session evaluations will be done by both participants and healthcare workers.

Do the intervention lead to adverse events? To what extent were individual goals met?

ELIGIBILITY:
Inclusion Criteria:

* both adults with and without disabilities recruited from different healthcare contexts.

Exclusion Criteria:

* Intellectual disability of the degree where the participant is not able to follow the protocol in Lev.

  * Insufficient command of the Swedish language/ unable to understand the content.
  * Severe psychiatric comorbidity that makes participation difficult (e.g. severe depression, severe suicidality, severe anxiety, ongoing psychosis, manic episode), other circumstances that could make participation hard (e.g. homelessness).

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion rate participants | within 3-4 months
  How many of the participants that started using Lev (i.e., completing screening with Lev-s) completed Lev (i.e., completing, 3 out of 4 session)

SECONDARY OUTCOMES:
Level of treatment credibility participants | Before and after taking part in Lev (after refers to completing the three sessions i.e, not including the booster session after three months). I.e within 6 weeks
  Was Lev perceived as creditable by participants using Treatment and Credibility Scale. Four items for credibility and one for expectation on a 10 point Likert scale where higher values indicate higher credibility.
Level of treatment credibility healthcare workers | Before and after taking part in Lev (after refers to completing the three sessions i.e, not including the booster session after three months)I.e within 6 weeks
  Was Lev perceived as creditable by healthcare workers using Treatment and Credibility Scale . Four items for credibility and one for expectation on a 10 point Likert scale where higher values indicate higher credibility.
Treatment satisfaction participants (individual sessions) | After completing the first session in Lev. An average of 1-2 weeks from baseline
  Treatment satisfaction will be evaluated after session 1 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  After the meeting today, my knowledge of how I can change my lifestyle have increased.
  I will benefit from what we talked about during the meeting today The content of the meeting felt relevant based on my own experiences I understood the advice and strategies I was given that will help my change mine lifestyle habits I feel confident in how to use the advice and strategies I will use the advice and strategies I was listened to, the therapist understood my situation I was involved and helped to come up with suggestions for how I can reach my goals Is there something else you would like to add?
Treatment satisfaction participants (individual sessions) | After completing the second session in Lev. An average of 2-3 weeks from baseline
  Treatment satisfaction will be evaluated after session 2 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  After the meeting today, my knowledge of how I can change my lifestyle have increased.
  I will benefit from what we talked about during the meeting today The content of the meeting felt relevant based on my own experiences I understood the advice and strategies I was given that will help my change mine lifestyle habits I feel confident in how to use the advice and strategies I will use the advice and strategies I was listened to, the therapist understood my situation I was involved and helped to come up with suggestions for how I can reach my goals Is there something else you would like to add?
Treatment satisfaction participants (individual sessions) | After completing the third session in Lev. An average of 3-4 weeks from baseline
  Treatment satisfaction will be evaluated after session 3 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  After the meeting today, my knowledge of how I can change my lifestyle have increased.
  I will benefit from what we talked about during the meeting today The content of the meeting felt relevant based on my own experiences I understood the advice and strategies I was given that will help my change mine lifestyle habits I feel confident in how to use the advice and strategies I will use the advice and strategies I was listened to, the therapist understood my situation I was involved and helped to come up with suggestions for how I can reach my goals Is there something else you would like to add?
Treatment satisfaction participants (individual sessions) | After completing the booster session in Lev. An average of 3-4 month from baseline
  Treatment satisfaction will be evaluated after booster session using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  After the meeting today, my knowledge of how I can change my lifestyle have increased.
  I will benefit from what we talked about during the meeting today The content of the meeting felt relevant based on my own experiences I understood the advice and strategies I was given that will help my change mine lifestyle habits I feel confident in how to use the advice and strategies I will use the advice and strategies I was listened to, the therapist understood my situation I was involved and helped to come up with suggestions for how I can reach my goals Is there something else you would like to add?
Treatment satisfaction participants (the three sessions) | Directly after completing the last treatment module in LEV (approximately at 3-4 weeks from baseline)]
  Treatment satisfaction will be evaluated after competing the three sessions using Patient Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  As a whole, the Lev has been clearly focused on how I can live healthier My knowledge of how I can have healthier habits has increased I can better deal with problems connected to my health-related habits I have had the opportunity to contribute opinions during the Lev I would consider participating in a similar interventions in the future The participants also rated the course as a whole following the school grading system ''Failed,'' ''Passed,'' ''Passed with distinction,'' and ''Passed with special
Treatment satisfaction participants (the whole intervention including the booster session) | Directly after completing the last treatment module in LEV (approximately at 3-4 month from baseline)]
  Treatment satisfaction will be evaluated after competing the whole intervention using Patient Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  As a whole, the Lev has been clearly focused on how I can live healthier My knowledge of how I can have healthier habits has increased I can better deal with problems connected to my health-related habits I have had the opportunity to contribute opinions during the Lev I would consider participating in a similar interventions in the future The participants also rated the course as a whole following the school grading system ''Failed,'' ''Passed,'' ''Passed with distinction,'' and ''Passed with special
Open answer questions regarding Treatment satisfaction measured by The Evaluation Questionnaire for participants | Directly after completing the third session in LEV (approximately at 3-4 weeks from baseline)]
  The treatment satisfaction questionnaire also included open questions that will be analyses using a qualitative thematic approach including the following questions:
  I feel that participating in Lev helped me in these ways How could the Lev have been better? What could I have done differently myself? Is there anything else you would like to add? A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.
  I would consider participating in a similar interventions in the future The participants also rated the course as a whole following the school grading system ''Failed,'' ''Passed,'' ''Passed with distinction,'' and ''Passed with special
Open answer questions regarding Treatment satisfaction measured by The Evaluation Questionnaire for participants | Directly after completing the booster session in LEV (approximately at 3-4 month from baseline)]
  The treatment satisfaction questionnaire also included open questions that will be analyses using a qualitative thematic approach including the following questions:
  I feel that participating in Lev helped me in these ways How could the Lev have been better? What could I have done differently myself? Is there anything else you would like to add? A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.
  I would consider participating in a similar interventions in the future.
  The participants also rated the course as a whole following the school grading system ''Failed,'' ''Passed,'' ''Passed with distinction,'' and ''Passed with special
Treatment satisfaction healthcare workers (individual sessions) | After completing the first session in Lev. An average of 1-2 weeks from baseline
  Treatment satisfaction will be evaluated after session 1 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  The content of this session feels relevant The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist Is there something else you would like to add?
Treatment satisfaction healthcare workers (individual sessions) | After completing the first session in Lev. An average of 2-3 weeks from baseline
  Treatment satisfaction will be evaluated after session 2 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  The content of this session feels relevant The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist Is there something else you would like to add?
Treatment satisfaction healthcare workers (individual sessions) | After completing the first session in Lev. An average of 3-4 weeks from baseline
  Treatment satisfaction will be evaluated after session 3 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  The content of this session feels relevant The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist Is there something else you would like to add?
Treatment satisfaction healthcare workers (individual sessions) | After completing the first session in Lev. An average of 3-4 months from baseline
  Treatment satisfaction will be evaluated after the booster session using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  The content of this session feels relevant The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist Is there something else you would like to add?
Well-being before and after the intervention measures by The Evaluation Questionnaire | Directly after completing the third treatment module in LEV (approximately at 3-4 weeks)
  ("How would you rate your well-being prior to the intervention?", "How would you rate your current well-being") at T1 and T2 on a scale 1-10 (1= very poor, 10= very good)
Well-being before and after the intervention measures by The Evaluation Questionnaire | Directly after completing the booster session module in LEV (approximately at 3-4 months)
  ("How would you rate your well-being prior to the intervention?", "How would you rate your current well-being") at T1 and T2 on a scale 1-10 (1= very poor, 10= very good)
Adverse events after the intervention | During the intervention up to week approximately 3-4 months
  Adverse events will be defined as spontaneous oral complaints or instances when patients stated that they experienced negative or unwanted effects during the intervention period.
  Serious adverse events will be defined as events that involved hospital care/hospitalization, etc. due to the intervention.
To what extent were individual goals met? | Directly after completing the third treatment module in LEV (approximately at 3-4 weeks)
  The healthcare worker assesses to what extent the goals have been met using the goal attainment scale. 5 point scale where high vales indicate that goals have been reached to a higher extent.
To what extent were individual goals met? | Directly after completing the booster session module in LEV (approximately at 3-4 months)
  The healthcare worker assesses to what extent the goals have been met using the goal attainment scale. 5 point scale where high vales indicate that goals have been reached to a higher extent.
Self-efficacy for promoting health behaviors for their children | Directly after completing the third session in LEV (approximately at 3-4 weeks)
  Participants are asked to assess self-efficacy for promoting health behaviors using the "Parental self-efficacy for healthy dietary and physical activity behaviors in preschool children (PDAP) including 24 items on a 0-10 point scale where high values indicate higher self-efficacy
Self-efficacy for promoting health behaviors for their children | Directly after completing the booster session in LEV (approximately at 3-4 month)
  Participants are asked to assess self-efficacy for promoting health behaviors using the "Parental self-efficacy for healthy dietary and physical activity behaviors in preschool children (PDAP) including 24 items on a 0-10 point scale where high values indicate higher self-efficacy
Do Lev lead to healthier habits? | Before and after taking part in Lev (after is after the third, 3-4 weeks, as wells as after the booster session, 3-4 month)
  The Lev-s will be used to measure diet and physical activity before and after taking part in Lev. The scale includes 4 levels where higher levels indicate healthier habits.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sjöwall, PhD, Principal Investigator — Region Stockholm
Locations (1):
- Region Stockholm, Stockholm, Stockholm, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No
Douglas Sjöwall will be responsible for granting access to data only to researchers who are participating in the publications